CLINICAL TRIAL: NCT05967351
Title: A Phase 3, Multinational, Long-term Follow-up Study to Evaluate Safety and Efficacy in Subjects Who Have Previously Received SRP-9001 in a Clinical Study
Brief Title: A Long-term Follow-up Study of Participants Who Received Delandistrogene Moxeparvovec (SRP-9001) in a Previous Clinical Study
Acronym: EXPEDITION
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRP-9001-305; 2023-505043-39-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Pediatric; Long-term; Follow-up; Safety; Efficacy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Delandistrogene Moxeparvovec (Experimental): Participants received delandistrogene moxeparvovec in a previous clinical study.
  Interventions: Genetic: delandistrogene moxeparvovec

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — No study drug will be administered as part of this study. Eligible participants who received treatment with delandistrogene moxeparvovec during a previous clinical study will be included.
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS

SUMMARY:
The purpose of this study is to provide a single clinical study with a uniform approach to monitoring long-term safety and efficacy in participants who received delandistrogene moxeparvovec in a previous clinical study. No study drug will be administered as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Received delandistrogene moxeparvovec for Duchenne muscular dystrophy in a previous clinical study.
* Has (a) parent(s) or legal caregiver(s) or is ≥18 years of age and able to understand and comply with the study visit schedule and all other protocol requirements.

Exclusion Criteria:

* Not applicable

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2033-10-31 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Treatment-emergent Adverse Event (TEAE), Serious Adverse Event (SAE), and Adverse Event of Special Interest (AESI) | Up to 10 years

SECONDARY OUTCOMES:
Change in the North Star Ambulatory Assessment (NSAA) Total Score From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in Time to Rise From Floor From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in the Time of 10-meter Walk/Run (10MWR) From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in Performance of Upper Limb (PUL) (Version 2.0) Total Scores From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in PUL (Version 2.0) Domain Specific Scores From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in Forced Vital Capacity Percent (FVC%) Predicted From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in Peak Expiratory Flow Percent (PEF%) Predicted From Pre-infusion Baseline to the End of the Study Participation of Delandistrogene Moxeparvovec | Baseline, up to 10 years
Change in Cardiac Magnetic Resonance Imaging (MRI) Findings From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years
Change in Musculoskeletal MRI Findings From Pre-infusion Baseline of Delandistrogene Moxeparvovec to the End of the Study Participation | Baseline, up to 10 years

CONTACTS AND LOCATIONS:
Locations (38):
- United States (22):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford (LPCH), Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa ICTS Clinical Research Unit, Iowa City, Iowa
  - The Johns Hopkins Hospital, Rubenstein Child Health Bldg, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Pediatric Neuromuscular Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Lenox Baker Children's Hospital (Duke University), Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Chiildren's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Health Specialty Center, Dallas, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital Wisconsin, Milwaukee, Wisconsin
- Universitair Ziekenhuis Gent, Neuromuscular Reference Centre (NMRC), Ghent, East Flanders, Belgium
- Universitätsklinikum Essen - Klinik für Kinderheilkunde I, Essen, North Rhine-Westphalia, Germany
- Hong Kong Children's Hospital, Hong Kong, Hong Kong
- Italy (3):
  - UOC Neurologia Pediatrica e Malattie Muscolari, Istituto G. Gaslini, Istituto Pediatrico di Ricovero e Cura a Carattere Scientifico, Genova
  - UOC Neurologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - UOC Neuropsichiatria Infantile, Area Salute del Bambino, Fondazione Policlinico Universitario A. Gemelli IRCCS, Universita Cattoclica del Sacro Cuore, Roma
- Japan (3):
  - Kobe University Hospital, Kobe, Hyōgo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario y Politecnico La fe. Neurology Department, Valencia
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Institute of Translational and Clinical Research, Newcastle upon Tyne